CLINICAL TRIAL: NCT02611232
Title: Incretin-based Therapy in Preclinical Type 1 Diabetes in Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Riitta Veijola, Professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LiraAAB18-30; 2014-003667-37 (EudraCT Number); 3-SRA-2014-301-M-R (Other Grant/Funding Number: Juvenile Diabetes Research Foundation International); U1111-1176-6062 (Other: WHO)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Type 1; Diabetes, Insulin-Dependent; Liraglutide; Preclinical Type 1 Diabetes; GLP-1 Analogue
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Victoza® (Active Comparator): Subjects with preclinical type 1 diabetes aged 18-30 years are treated with Victoza® (liraglutide)
  Interventions: Drug: Victoza®
- Placebo (Placebo Comparator): Subjects with preclinical type 1 diabetes aged 18-30 years are treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Victoza® — Daily subcutaneous injections with increasing doses up to 1.8 mg per day. Duration of treatment 6 months. Duration of follow-up 24 months.
  Arms: Victoza®
Drug: Placebo — Daily subcutaneous injections with increasing doses up to 1.8 mg per day. Duration of treatment 6 months. Duration of follow-up 24 months.
  Arms: Placebo

SUMMARY:
The main objectives of the trial are to study whether daily treatment with liraglutide improves insulin secretion and glucose metabolism, and whether liraglutide treatment is tolerable and safe in subjects with preclinical type 1 diabetes aged 18-30 years.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* positive for at least 2 biochemical islet autoantibodies
* have normal glucose tolerance in OGTT
* are not pregnant

Exclusion Criteria:

* allergic to liraglutide or other ingredients of Victoza®
* Type 1 diabetes
* diabetic ketoacidosis
* previous treatment in the last three months with any antidiabetic medication
* impaired liver or kidney function or on dialysis
* severe heart failure
* severe stomach or gut problem resulting in gastroparesis, or inflammatory bowel disease
* past or current history of pancreatitis
* serum calcitonin value above normal (>50 ng/l or ≥3.4pmol/l)
* presence of any chronic metabolic, hematologic or malignant disease
* obesity BMI ≥30
* pregnant females and females of childbearing potential who are not using adequate contraceptive methods.
* breast-feeding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
FPIR (first phase insulin response) | From baseline to 26 and 104 weeks
  First phase insulin response during 10-min IVGTT (intravenous glucose tolerance test )

SECONDARY OUTCOMES:
Safety: serum and urine amylase, serum lipase, serum calcitonin, hypoglycemia | From baseline to 26 and 104 weeks
  Safety: serum and urine amylase, serum lipase, serum calcitonin, hypoglycemia
Tolerability | From baseline to 26 and 104 weeks
  Tolerability: frequency of side effects, particularly hypoglycaemia and gastrointestinal symptoms
Serum C-peptide AUC | From baseline to 26 and 104 weeks
  Serum C-peptide area under the curve (AUC) during 2-hour OGTT (oral glucose tolerance test)

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Veijola, MD, Principal Investigator — University of Oulu
Locations (3):
- Finland (3):
  - University of Oulu and Oulu University Hospital, Oulu
  - University of Tampere and Tampere University Hospital, Tampere
  - University of Turku and Turku University Hospital, Turku

REFERENCES:
- [Derived] Kero J, Koskenniemi JJ, Karsikas S, Pokka T, Lou O, Toppari J, Veijola R. INnoVative trial design for testing the Efficacy, Safety and Tolerability of 6-month treatment with incretin-based therapy to prevent type 1 DIAbetes in autoantibody positive participants: A protocol for three parallel double-blind, randomised controlled trials (INVESTDIA). Diabet Med. 2022 Oct;39(10):e14913. doi: 10.1111/dme.14913. Epub 2022 Jul 22. PMID 35797241